CLINICAL TRIAL: NCT04394546
Title: WATCHMAN FLX Versus NOAC for Embolic ProtectION in in the Management of Patients With Non-Valvular Atrial Fibrillation
Brief Title: CHAMPION-AF Clinical Trial
Acronym: CHAMPION-AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: S2437
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Stroke; Bleeding
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Hemorrhage | interventions — N(4)-oleylcytosine arabinoside

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Device Group (Experimental): Randomized to WATCHMAN FLX Left Atrial Appendage Closure Device
  Interventions: Device: WATCHMAN FLX LAAC Device
- Control Group (Active Comparator): Randomized to non-vitamin K oral anticoagulant (NOAC)
  Interventions: Drug: Non-Vitamin K Oral Anticoagulant

INTERVENTIONS:
Device: WATCHMAN FLX LAAC Device — WATCHMAN FLX LAAC Device Implantation
  Other Names: WATCHMAN FLX Left Atrial Appendage Closure Device
  Arms: Device Group
Drug: Non-Vitamin K Oral Anticoagulant — Initiation or continuation of a NOAC drug
  Other Names: NOAC
  Arms: Control Group

SUMMARY:
The primary objective of this study is to determine if left atrial appendage closure (LAAC) with the WATCHMAN FLX device is a reasonable alternative to non-vitamin K oral anticoagulants in patients with non-valvular atrial fibrillation.

DETAILED DESCRIPTION:
This study is a prospective, randomized, multi-center global investigation. Subjects will be randomized to either the WATCHMAN FLX Left Atrial Appendage Closure Device ("Device Group") or a commercially available non-vitamin K oral anticoagulant ("Control Group").

ELIGIBILITY:
Inclusion Criteria:

* The subject is of legal age to participate in the study per the laws of their respective geography
* The subject has documented non-valvular atrial fibrillation (i.e., atrial fibrillation in the absence of moderate or greater mitral stenosis or a mechanical heart valve)
* The subject has a calculated CHA2DS2-VASc (congestive heart failure, hypertension, age ≥ 75 years, diabetes mellitus, stroke or transient ischemic attack (TIA), vascular disease, age 65 to 74 years, sex category) score of 2 or greater for men and 3 or greater for women
* The subject is deemed to be suitable for the protocol-defined pharmacologic regimens in both the test and control arms
* The subject or legal representative is able to understand and willing to provide written informed consent to participate in the trial
* The subject is able and willing to return for required follow-up visits and examinations

Exclusion Criteria:

* Subjects who are currently enrolled in another investigational study, except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments
* The subject requires long-term anticoagulation therapy for reasons other than AF-related stroke risk reduction, for example due to an underlying hypercoagulable state (i.e., even if the device is implanted, the subjects would not be eligible to discontinue OAC due to other medical conditions requiring chronic OAC therapy)
* The subject is contraindicated or allergic to oral anticoagulation medication and/or aspirin
* The subject is indicated for chronic P2Y12 platelet inhibitor therapy
* The subject had or is planning to have any cardiac or non-cardiac intervention or surgical procedure within 30 days prior to or 60 days after implant (including, but not limited to: cardioversion, percutaneous coronary intervention (PCI), cardiac ablation, cataract surgery, etc.)
* The subject had a prior stroke (of any cause, whether ischemic or hemorrhagic) or transient ischemic attack (TIA) within the 30 days prior to enrollment
* The subject had a prior major bleeding event per ISTH definition within the 30 days prior to randomization. Lack of resolution of related clinical sequelae or planned and pending interventions to resolve bleeding/bleeding source, are a further exclusion regardless of timing of the bleeding event
* The subject has an active bleed
* The subject has a reversible cause of AF or transient AF
* The subject is absent of a left atrial appendage (LAA) or the LAA is surgically ligated
* The subject has had a myocardial infarction (MI) documented in the clinical record as either a non-ST elevation MI (NSTEMI) or as an ST-elevation MI (STEMI), with or without intervention, within 30 days prior to enrollment
* The subject has a history of atrial septal repair or has an atrial septal device (ASD)/patent foramen ovale (PFO) device
* The subject has an implanted mechanical valve prosthesis in any position
* The subject has a known contraindication to percutaneous catheterization procedure
* The subject has a known contraindication to transesophageal echo (TEE)
* The subject has a cardiac tumor
* The subject has signs/symptoms of acute or chronic pericarditis.
* The subject has an active infection
* There is evidence of tamponade physiology
* The subject has New York Heart Association Class IV Congestive Heart Failure at the time of enrollment
* The subject is of childbearing potential and is, or plans to become, pregnant during the time of the study (method of assessment upon study physician's discretion)
* The subject has a documented life expectancy of less than 3 years

Transthoracic Echo Exclusion Criteria:

* The subject has left ventricular ejection fraction ( LVEF) < 30%
* The subject has an existing pericardial effusion with a circumferential echo-free space > 5mm
* The subject has a high-risk PFO with an atrial septal aneurysm excursion > 15mm or length > 15mm
* The subject has significant mitral valve (MV) stenosis (i.e., MV area <1.5 cm2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
WATCHMAN FLX is non-inferior (NI) for the occurrence of stroke, cardiovascular death, and systemic embolism | 36-months
  non-inferiority
WATCHMAN FLX is superior for non-procedural bleeding (ISTH major bleeding and clinically relevant non-major bleeding) | 36-months
  superiority
WATCHMAN FLX is non-inferior (NI) for the occurrence of ischemic stroke and systemic embolism | 60-months
  non-inferiority

SECONDARY OUTCOMES:
The occurrence of ISTH major bleeding | 60-months
  superiority
The occurrence of cardiovascular (CV) death, all stroke, systemic embolism (SE), and non-procedural bleeding (ISTH major bleeding and clinically relevant non-major bleeding) | 60-months
  superiority
The occurrence of ISTH Major Bleeding | 36-months
  Non-Inferiority
The occurrence of cardiovascular (CV) death, all stroke, systemic embolism (SE), and non-procedural bleeding (ISTH major bleeding and clinically relevant non-major bleeding) | 36-months
  Non-inferiority

CONTACTS AND LOCATIONS:
Overall Officials: Marty Leon, MD, Study Chair — New York-Presbyterian Heart Valve Center/Columbia University Irving Medical Center; Kenneth A Ellenbogen, MD, Study Chair — Virginia Commonwealth University; Shephal Doshi, MD, Principal Investigator — Pacific Heart Institute and Providence St. John's Health Center; Saibal Kar, MD, Principal Investigator — HCA Healthhcare /Los Robles Health System
Locations (141):
- United States (95):
  - Grandview Medical Center, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Arrhythmia Research Center, Phoenix, Arizona
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Scottsdale Healthcare - Shea, Scottsdale, Arizona
  - Tucson Medical Center Healthcare, Tucson, Arizona
  - Arrythmia Research Group, Jonesboro, Arkansas
  - Sharp Chula Vista Medical Center, Chula Vista, California
  - Marin General Hospital, Greenbrae, California
  - Scripps Memorial Hospital, La Jolla, California
  - Los Robles Hospital and Medical Center, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Mercy General Hospital, Sacramento, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - St. John's Health Center, Santa Monica, California
  - Colorado Springs Cardiologist, P.C., Colorado Springs, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Christiana Hospital, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Manatee Memorial Hospital, Bradenton, Florida
  - Bay Area Cardiology Associates, P.A., Brandon, Florida
  - Broward General Medical Center, Fort Lauderdale, Florida
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Lakeland Regional Medical Center, Lakeland, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Community Hospital, Munster, Indiana
  - Mercy Hospital Medical Center, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Norton Hospital, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Lahey Clinic Hospital, Burlington, Massachusetts
  - Charlton Memorial, Fall River, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Sparrow Health System - Sparrow Hospital, Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Mayo Clinic Foundation, Rochester, Minnesota
  - Centracare Heart and Vascular Center, Saint Cloud, Minnesota
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Billings Clinic, Billings, Montana
  - Bergan Cardiology, Omaha, Nebraska
  - The Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Catholic Medical Center, Manchester, New Hampshire
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Kaleida Health, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Rochester General Hospital, Rochester, New York
  - St. Francis Hospital, Roslyn, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - OhioHealth Research and Innovation Institute-Riverside Methodist Hospital, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Legacy Emanuel Hospital & Health Center, Portland, Oregon
  - Pinnacle Health at Harrisburg Hospital, Harrisburg, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Trident Medical Center, Charleston, South Carolina
  - Medical University of South Carolina, Columbia, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Methodist Le Bonheur Healthcare, Germantown, Tennessee
  - Centennial Medical Center, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research, Austin, Texas
  - Heart Hospital of Austin, Austin, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Methodist Texsan Hospital, San Antonio, Texas
  - Christus Trinity Mother Frances Health System, Tyler, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Providence Regional Medical Center Everett, Everett, Washington
  - Swedish Medical Center, Seattle, Washington
  - CHI Franciscan Health System, Tacoma, Washington
  - PeaceHealth Southwest Medical, Vancouver, Washington
  - Monongalia General Hospital, Morgantown, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (3):
  - St. Vincent's Hospital-Sydney, Darlinghurst, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - Westmead Hospital, Bella Vista
- Belgium (2):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - CHU de Charleroi, Charleroi
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Institut universitaire de Cardiologie et de Pneumologie de Quebec, Québec
- Aarhus University Hospital, Aarhus, Denmark
- France (3):
  - Hopital Cardiologique de Lyon, Bron
  - CHU Grenoble-Hopital Michallon, Grenoble
  - Hospital de la Pitie-Salpetriere, Paris
- Germany (9):
  - Charite, Campus Benjamin Franklin, Berlin
  - SANA Kliniken Oberfranken Coburg GmbH, Coburg
  - Herzzentrum Dresden GmbH, Dresden
  - St.Johann Nepomuk Katholisches Hospitalvereinigung Thüringen GmbH, Erfurt
  - Elisabeth Krankenhaus Essen, Essen
  - St. Katharinen Krankenhaus, Frankfurt
  - Cardiologicum Hamburg Praxis Wandsbek, Hamburg
  - Universitaetsklinikum Schleswig-Holstein, Lübeck
  - Klinikum der Ludwig-Maximilians-Universitat, München
- Israel (2):
  - Shaare Zedek Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
- Italy (4):
  - Fondazione Toscana Gabriele Monasterio, Pisa, PI
  - Azienda Ospedaliera Careggi, Florence
  - Ospedale Degli Infermi, Rivoli
  - Instituto Clinico Humanitas, Rozzano
- Japan (10):
  - Chiba University Hospital, Chiba, Chiba
  - Kokura Memorial Hospital, Kitakyushu-shi, Fukuoka
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - Mitsui Memorial Hospital, Chiyoda-ku, Tokyo
  - Shonan Kamakura General Hospital, Okamoto
  - Kurashiki Central Hospital, Okayama
  - Toho University Ohashi Medical Center, Tokyo
  - Toyama University Hospital, Toyama
  - Toyohashi Heart Center, Toyohashi
  - University of Tsukuba Hospital, Tsukuba
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands
- Poznan University of Medical Sciences, Długa, Poznań, Poland
- King Fahed Medical City- Prince Salman Cardiac Center, Riyadh, Saudi Arabia
- Spain (3):
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital de Leon, León
  - Hospital Clinico Salamanca, Salamanca
- University Hospital Zurich, Zurich, Switzerland
- United Kingdom (3):
  - Royal Sussex County Hospital, Brighton
  - Glenfield Hospital, Leicester
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
URL: http://www.bostonscientific.com/content/gwc/en-US/data-sharing-requests.html

REFERENCES:
- [Derived] Kar S, Doshi SK, Alkhouli M, Camm AJ, Coylewright M, Gibson MC, Granger CB, Gurol ME, Huber K, Mansour M, Nair DG, Natale A, Pocock SJ, Reddy VR, Saliba W, Christen T, Allocco DJ, Ellenbogen KA, Leon MB. Rationale and design of a randomized study comparing the Watchman FLX device to DOACs in patients with atrial fibrillation. Am Heart J. 2023 Oct;264:123-132. doi: 10.1016/j.ahj.2023.05.022. Epub 2023 Jun 4. PMID 37279840